CLINICAL TRIAL: NCT02386488
Title: A Randomised, Open-label, Single-centre, Single- and Multiple-dose Interventional Study Investigating the Pharmacokinetic Properties of Vortioxetine in Healthy Young Chinese Men and Women
Brief Title: Pharmacokinetic Properties of Vortioxetine in Healthy Young Chinese Men and Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16060A
Record Dates: First submitted 2015-03-05; First posted 2015-03-12 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Vortioxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vortioxetine 10 mg single dose (Experimental): 8 men and 8 women
  Interventions: Drug: Vortioxetine 10 mg single dose
- Vortioxetine 20 mg single dose (Experimental): 8 men and 8 women
  Interventions: Drug: Vortioxetine 20 mg single dose
- Vortioxetine 10 mg multiple dose (Experimental): 8 men and 8 women
  Interventions: Drug: Vortioxetine 10 mg multiple dose
- Vortioxetine 20 mg multiple dose (Experimental): 8 men and 8 women
  Interventions: Drug: Vortioxetine 20 mg multiple dose

INTERVENTIONS:
Drug: Vortioxetine 10 mg single dose — 10 mg tablet for oral use, single dose
  Other Names: Lu AA21004
  Arms: Vortioxetine 10 mg single dose
Drug: Vortioxetine 20 mg single dose — Two 10 mg tablets for oral use, single dose,
  Other Names: Lu AA21004
  Arms: Vortioxetine 20 mg single dose
Drug: Vortioxetine 10 mg multiple dose — 10 mg tablet for oral use once, daily for 14 days.
  Other Names: Lu AA21004
  Arms: Vortioxetine 10 mg multiple dose
Drug: Vortioxetine 20 mg multiple dose — Two 10 mg tablets for oral use, once daily for 14 days.
  Other Names: Lu AA21004
  Arms: Vortioxetine 20 mg multiple dose

SUMMARY:
The purpose of this study is to determine the pharmacokinetic (PK) parameters of vortioxetine after single and multiple oral dosing to healthy Chinese men and women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young Chinese men or women
* Between 18 and 45 years of age (extremes included)
* BMI between 18.5 and 24 kg/m2 (extremes included)
* Body weight ≥45 kg.

Exclusion Criteria:

* Pregnant or lactating.
* Previously been dosed with vortioxetine
* The subject has taken any investigational medicinal products within 3 months prior to the first dose of IMP (investigational medicinal product)

Other protocol defined inclusion and exclusion criteria may apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of vortioxetine and its metabolites: Cmax, AUC, t1/2, oral clearance, apparent volume of distribution, accumulation index, metabolic ratio | Day 1 to 312 hours post-dose
  Composite pharmacokinetic outcome measures (PK parameters: Cmax, AUC, t1/2, oral clearance, apparent volume of distribution, accumulation index, metabolic ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- CB801, Chengdu, China